CLINICAL TRIAL: NCT06569472
Title: Clinical Study of CD19 Targeting Chimeric Antigen Receptor T Lymphocytes (CAR-T) in the Treatment of Refractory Juvenile Dermatomyositis (RJDM)
Brief Title: Clinical Trial of CD19-targeted CAR-T Therapy for Refractory Juvenile Dermatomyositis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC068
Record Dates: First submitted 2024-08-21; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-07

CONDITIONS: Juvenile Dermatomyositis
Keywords: CAR-T; CD19
MeSH Terms: conditions — Dermatomyositis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19-targeted CAR-T (Experimental): The experiment was divided into two phases: dose exploration (Part A) and dose extension (Part B).
  Interventions: Biological: CD19-targetd CAR-T

INTERVENTIONS:
Biological: CD19-targetd CAR-T — Subjects underwent lymphocyte clearance chemotherapy and then received a single intravenous cell infusion

SUMMARY:
This is a Phase I clinical trial to evaluate the efficacy and safety of CD19-targeted CAR-T in the treatment of refractory juvenile dermatomyositis (RJDM).The experiment was divided into two phases: dose exploration (Part A) and dose extension (Part B).

DETAILED DESCRIPTION:
juvenile dermatomyositis (JDM) is a non-suppurative chronic autoimmune disease and the most common type of juvenile idiopathic inflammatory myopathy.Despite the active treatment measures, some JDM patients are still intolerant or unresponsive to the treatment, resulting in a high disability and mortality rate.Because CD19 is widely expressed on the surface of B lymphocytes, CD19 CAR-T can also cause deep depletion of other CD19+ B cells while killing cancer cells, which is expected to achieve immune reconstruction in patients with autoimmune diseases, and completely change the status quo that such patients need to take hormones and immunosuppressants for a long time.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥5 years and <17 years old
2. To meet the diagnostic criteria of JDM, four or five of the following criteria must be met:① symmetrical proximal muscle weakness; ②Characteristic skin changes, including positive dermatitis (purplish red rash on upper eyelid with periorbital edema) and Gottron papules (red patchy squamous papules on the back of knuckles); ③ The level of one muscle enzyme in serum was increased; ④ Positive myositis antibody; ⑤Electromyography shows denervation and myopathy; ⑥ Muscle biopsies showed necrosis and inflammation.
3. The classification criteria of RJDM must meet ① and any of the criteria②-④: ① Patients who are intolerant or unresponsive to glucocorticoids and at least 2 immunosuppressants, adequate hormone therapy and duration of at least 6 months; ② The disease progresses rapidly and/or involves organs such as lungs, heart and gastrointestinal tract; ③ Calcification of subcutaneous or muscle and joint tissues; ④ Repeated rashes or skin ulcers.
4. myositis specific antibody positive, defined as MDA-5, NXP2, TIF-1γ, Ro-52 and any other positive;
5. If the patient has SRP or HMGCR antibody positive immune-mediated necrotizing myopathy equivalent to RJDM, the inclusion criteria of (2) - (4) can be met.
6. The functions of important organs are basically normal:

   ① Cardiac function: left ventricular ejection fraction (LVEF) ≥55%, no obvious abnormality in electrocardiogram;

   ② Renal function: eGFR≥30ML/min/1.73m2;

   ③ Liver function: AST and ALT≤3.0 ULN, total bilirubin ≤2.0×ULN;

   ④ Lung function: Lung function is basically normal, SpO2≥92%;
7. Have the criteria for simple or intravenous blood collection, and no other contraindications for cell collection;
8. The subject of childbearing age has a negative urine pregnancy test result and agrees to take effective contraceptive measures during the test period until 1 year after the infusion;
9. The patient or his/her guardian agrees to participate in this clinical trial and signs an informed consent indicating that he/she understands the purpose and procedure of this clinical trial and is willing to participate in the study.

Exclusion Criteria:

1. Had previously received CAR T cell therapy;
2. Have other autoimmune or rheumatic diseases other than JDM;
3. primary immunodeficiency or severe secondary immunodeficiency that has not been corrected;
4. accompanied by serious infectious diseases, including but not limited to active tuberculosis, latent tuberculosis infection, active viral hepatitis, etc.;
5. Evidence of active malignant disease or diagnosis of malignant tumor (including hematological malignancies and solid tumors, except resected and cured skin basal cell carcinoma)
6. Congenital heart disease or history of acute myocardial infarction within 6 months before screening, or severe arrhythmias (including multi-source frequent supraventricular tachycardia, ventricular tachycardia, etc.); Or combined with a large number of pericardial effusion, serious myocarditis, etc.; Or patients with unstable vital signs who need hypertensive drugs to maintain their blood pressure;
7. suffering from other diseases that require long-term use of glucocorticoids or immunosuppressants;
8. There is an active or uncontrollable infection that requires systemic treatment within 1 week prior to screening;
9. Received solid organ transplantation or hematopoietic stem cell transplantation within 3 months before screening; Acute graft-versus-host disease (GVHD) of grade 2 or above was present within 2 weeks prior to screening;
10. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer greater than the normal reference value range; Or hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA titer greater than the normal reference value range; Or positive for human immunodeficiency virus (HIV) antibodies; Or syphilis test positive; Or cytomegalovirus (CMV) DNA test positive;
11. Had received live vaccine within 4 weeks prior to screening;
12. Positive blood pregnancy test;
13. Patients with known malignant diseases such as tumors before screening;
14. Patients who had participated in other clinical trials within 3 months prior to enrollment;
15. Situations in which other investigators consider it inappropriate to participate in the study.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of CAR-T in the treatment of refractory juvenile dermatomyositis [Safety and Tolerability] | 28 days
  The incidence of adverse events after CAR-T cell infusion was assessed by the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 5.0).including the type, frequency and severity of adverse events
To evaluate the efficacy of CAR-T in the treatment of refractory juvenile dermatomyositis [Effectiveness] | 2month,3months
  Disease improvement rate: The number of subjects who achieved disease improvement as a percentage of all subjects who received transfusions.
Duration of Response (DOR) of CAR-T treatment in the treatment of refractory juvenile dermatomyositis [Effectiveness] | 2 years
  DOR will be assessed from the first assessment of remission to the first assessment of recurrence or progression of the disease or death from any cause

SECONDARY OUTCOMES:
AUCS of CD19 CAR-T cells [Cell dynamics] | 3 months
  AUCS is defined as the area under the curve in 90 days
CMAX of CD19 CAR-T cells [Cell dynamics] | 3 months
  CMAX is defined as the highest concentration of CEA CAR-T cells expanded in peripheral blood
TMAX of CD19 CAR-T cells[Cell dynamics] | 3 months
  TMAX is defined as the time to reach the highest concentration

OTHER OUTCOMES:
To evaluate the effects of CD19-targeting CAR T cell preparations on the weight of children | 2 years
  Weight in kilograms were monitored after transfusion until subjects reached 18 years of age
To evaluate the effects of CD19-targeting CAR T cell preparations on the height of children | 2 years
  Height in meters were monitored after transfusion until subjects reached 18 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Meiping Lu, M.D, Principal Investigator — Children's Hospital, Zhejiang University School of Medicine
Locations (1):
- Children's Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China